CLINICAL TRIAL: NCT06355973
Title: A Pilot Study for Efficacy of Cognitive and Physical Training in Patients With Mild Cognitive Impairment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MinYoung Kim, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, MinYoung Kim, MD, PhD, Sponsor-Investigator, Bundang CHA Hospital
Organization: Bundang CHA Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-01-061
Record Dates: First submitted 2024-03-19; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Patients With Mild Cognitive Impairment (MCI)

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Using tablets and workbooks. (Experimental): Using tablets and workbooks Cognitive and physical function training self-programming for 6 weeks.
  Interventions: Device: Using tablets and workbooks cognitive function.; Device: self-programming of physical function training.
- Only self-programming of physical function training. (Experimental): Only self-programming of physical function training is provided Implemented for 6 weeks.
  Interventions: Device: self-programming of physical function training.

INTERVENTIONS:
Device: Using tablets and workbooks cognitive function. — Cognitive training programs corresponding to memory, attention, time and space, and orientation are conducted for 35 to 60 minutes.
  Arms: Using tablets and workbooks.
Device: self-programming of physical function training. — The fitness program consisting of stretching, muscle strength, coordination, and aerobic exercise lasts 20 to 30 minutes, and additional 3-4 times/mainly 30 to 40 minutes of aerobic exercise.

SUMMARY:
This is to find out the effectiveness of cognitive and physical function training for patients with mild cognitive impairment.

It is for the prevention and treatment of dementia in the future. randomized, Pilot Study.

ELIGIBILITY:
Inclusion Criteria:

1. men and women aged 60 or older
2. A person who falls within the abnormal range of the Montreal Cognitive Assessment (MoCA) test
3. a person who can independently carry out daily life
4. If the subject or legal representative voluntarily decides to participate and agrees in writing to comply with the precautions after hearing and fully understanding the detailed explanation of this clinical study

Exclusion Criteria:

1. A person diagnosed with Alzheimer's dementia or other causes (stroke, brain tumor, cerebral palsy, dementia, Parkinson's disease, etc.)
2. A person with unstable cardiovascular system, digestive system, respiratory system, endocrine system, etc. and poor general condition
3. Patients who have participated in other treatment clinical studies or who have participated in other treatment clinical studies within the last 30 days
4. Other cases where the researcher determines that participation in this clinical study is not appropriate

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) | screening - 6 weeks - 3 months
  K-MoCA is a measure of memory loss or other symptoms of cognitive decline. It includes 30 questions and a task that takes about 12 minutes to complete. The score can range from 0 to 30. A score of 26 or higher is considered normal.

SECONDARY OUTCOMES:
Korean-Mini Mental Status Examination (K-MMSE) | Baseline - 6 weeks - 3months
  K-MMSE is a measurement of cognitive level. Any score of 24 or more (out of 30) indicates a normal cognition. Below this, scores can indicate severe(≤9 points), moderate (10-18 points) or mild (19-23 points) cognitive impairment. The raw score may also need to be corrected for educational attainment and age.
Clinical Dementia Rating (CDR) | Baseline - 3months
  CDR is a rating scale for staging patients diagnosed with dementia. The CDR evaluates cognitive, behavioral and functional aspects of Alzheimer disease and other dementias. It is calculated on the basis of testing six different cognitive and behavioral domains such as memory, orientation, judgment and problem solving, community affairs, home and hobbies performance, and personal care. The CDR is based on a scale of 0-3: no dementia (CDR = 0), questionable dementia (CDR = 0.5), MCI (CDR = 1), moderate cognitive impairment (CDR = 2) and severe cognitive impairment (CDR = 3)
Clinical Global Impressions of Change (CGIC) | Baseline - 6 weeks- 3months
  CGIC is a commonly used measure to measure the severity, treatment rate, and treatment effectiveness of symptoms in the treatment process or research of patients with mental illness.
Instrumental Activities of Daily Living (I-ADL) | Baseline - 6 weeks- 3months
  I-ADL consists of skills and behaviors necessary for social life such as "money management," "households," "phone use," and "drugs," and helps evaluate the degree of social and professional functioning of the elderly with dementia.
Berg Balance Scale (BBS) | Baseline - 6 weeks- 3months
  BBS is a measurement of balancing function. A five-point ordinal scale, ranging from 0-4. "0" indicates the lowest level of function and "4" the highest level of function. Total score = 56
Geriatric Quality of Life-Dementia (GQOL-D) | Baseline - 6 weeks- 3months
  GQOL-D is a tool for evaluating the quality of life of the elderly with dementia and consists of a four-point scale of 15 items, including 13 items that measure physical health, psychological health, social relationships and environment, and two items that measure overall health and life satisfaction.
Geriatric Depression Scale (GDSd) | Baseline - 6 weeks- 3months
  GDS is a 30-item self-report assessment used to identify depression in the elderly. One point is assigned to each answer and the cumulative score is rated on a scoring grid. The grid sets a range of 0-9 as "normal", "10-19" as "mildly depressed", and 20-30 as "severely depressed".
Global Deterioration Scale (GDS) | Baseline - 3months
  GDS is one of the representative rating scales that suggests the severity of dementia patients and is used as a useful test tool for clinical trials of dementia treatments and early diagnosis of dementia.
Electroencephalography | Baseline - 6 weeks- 3months
  EEG is a measurement of electrical activity in the brain using small electrodes attached to the scalp for diagnose brain disorders.

CONTACTS AND LOCATIONS:
Overall Officials: MinYoung Kim, MD, PhD, Principal Investigator — CHA Bundang Medical Center